CLINICAL TRIAL: NCT05235503
Title: Influence of Δ9-tetrahydrocannabinol (THC) on Oxycodone Induced Ventilatory Depression in Healthy Volunteers
Acronym: COXY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, Coordinating investigator, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: P21.030; 2021-000083-29 (EudraCT Number); NL76443.058.21 (Other: CCMO Netherlands)
Record Dates: First submitted 2021-11-30; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Depression; Cannabis Use; Opioid Use
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Medical Marijuana

STUDY DESIGN:
Intervention Model Description: Double blind, randomized cross-over, placebo-controlled design.
Who Masked: Participant, Investigator
Masking Description: Blinding via pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20mg Oxycodon (capsule) + 100 mg Bedrocan (vaporized) (Experimental): As stated above
  Interventions: Drug: Medicinal cannabis in combination with oxycodon
- Placebo oxycodon (capsule) + 100 mg Bedrocan (vaporized) (Placebo Comparator): As stated above
  Interventions: Drug: Medicinal cannabis in combination with placebo oxycodon

INTERVENTIONS:
Drug: Medicinal cannabis in combination with oxycodon — The intervention will be administering the combination of medicinal cannabis in combination with oxycodon
  Arms: 20mg Oxycodon (capsule) + 100 mg Bedrocan (vaporized)
Drug: Medicinal cannabis in combination with placebo oxycodon — The intervention will be administering the combination of medicinal cannabis in combination with placebo oxycodon
  Arms: Placebo oxycodon (capsule) + 100 mg Bedrocan (vaporized)

SUMMARY:
Rationale:

Opioid misuse and abuse are common problems in the Western world. The rate of unintentional drug overdose is rapidly increasing, not only in the Unites States but also in the Netherlands. Additionally, it is well known that opioids are often used (and abused) in combination with other legal or illicit substances, for example cannabis, including medicinal (i.e. doctor prescribed) cannabis. A major opioid-induced adverse effect is respiratory depression and there are no data that show how oxycodone interacts with cannabis on the ventilatory control system. An appreciable effect is possible given the sedative effects of cannabis. Moreover, investigators previously showed that combining even a low dose of oxycodone (20 mg) with ethanol increased the likelihood of an apneic event (van der Schrier et al. Anesthesiology 2017; 102: 115-122). Because of this side effect and also due to the rising number of addicted chronic opioid users, there is an increasing imminent societal, political and medical interest in advancing research on opioids, opioid-drug interaction and alternatives for the treatment of various chronic illnesses and chronic pain.

Hypothesis: The investigators hypothesize that cannabis will amplify the ventilatory depressant effect of oxycodone (primary end-point).

Objective: The objective of the study is to quantify the interactive effect of Δ9-tetrahydrocannabinol (THC) and oxycodone on ventilatory control.

Study design: Double blind, randomized cross-over, placebo-controlled design.

Study population: Healthy human volunteers between the age of 18 and 45 years old.

Intervention:

Visit A: placebo capsule at t = 0 min + Bedrocan (22.4 mg THC) at t = 90 and 270 min; Visit B: oxycodone 20 mg at t = 0 min + Bedrocan (22.4 mg THC) at t = 90 and 270 min.

Main study parameters/endpoints:

Primary endpoint: The effect of inhaled THC on ventilation at an end-tidal PCO2 = 55 mmHg without and with concomitant intake of 20 mg oxycodone immediate release (IR) capsule in healthy volunteers 120 min after oxycodone intake.

Secondary endpoints: (1) Outcome of Bowdle and Bond & Lader questionnaires; (2) Level of sedation; (3) Pain Pressure Threshold; (4) slope of the hypercapnic ventilatory response; (5) plasma concentrations of THC, 11-OH-THC and oxycodone; a secondary analysis will be performed on the pharmacokinetic and pharmacodynamic data (PKPD modeling).

DETAILED DESCRIPTION:
General study design The design of the study is randomized, placebo-controlled crossover. Each subject will be studied twice, on one occasion he or she will receive THC and a placebo opioid capsule, and on the other occasion THC and an oxycodone capsule. The visits to the lab will be randomized, the washout period between the two occasions is at least 10 days. Subjects will be evaluated by a physician at screening and only healthy volunteers, aged 18-45 years, with a body mass index < 30 kg.m-2, are eligible to participate in the study.

Upon arrival in the laboratory (K5-120), the investigators will perform a urinary drug test and breath alcohol test. When these tests are positive, the subject is excluded from further participation. A venous and an arterial line will be placed. The venous line is used for fluid administration (NaCl/Glucose 50-100 ml/h), the arterial line is for blood sample drawing.

Next, the first hypercapnic ventilatory responses (HCVR) will be obtained (t = -30 min). This is the pre-drug baseline measurement. At t = 0, the subjects will receive 20 mg oxycodone immediate release or placebo. Next, the investigators will obtain HCVRs at 1-hour intervals until 6 hours after oxycodone/placebo intake. At t = 1.5 h and at t = 4.5 h the subject will inhale 100 mg Bedrocan. Breathing will be measured using the "dynamic end-tidal forcing" (DEF) system. At specific time points the investigators will draw 10 mL blood for measurement of drug concentrations. After 8 hours of measurement, we will assess whether the HCVR is still depressed. If so, the investigators will take another measurement at t = 9 h and reassess the HCVR. If still depressed, a last response will be obtained at t = 10 h. If necessary, the subject will stay overnight in the hospital. This will be decided by the physician-investigator. For example, the subject may still be sedated.

The hypercapnic ventilatory response To obtain the HCVR curve, the subject will rebreathe a gas mixture from a 6 L rebreathing balloon bag containing 7% carbon dioxide in 93% oxygen. The slope of the response and ventilation at 55 mmHg will be used in the analysis.

Oxycodone intake:

At t = 0, the subject will ingest 1 oxycodone 20 mg immediate release or a placebo capsule with 100 mL water. Both drugs will be obtained from the LUMC pharmacy.

Cannabis inhalation: Bedrocan is vaporized using the CE-marked Volcano Medic vaporizer (Storz & Bickel GmbH & Co, Tuttlingen, Germany), a safe and reliable method of intrapulmonary administration of cannabinoids. The Volcano heats the homogenized plant material to 210 °C to allow for conversion of the THC acid and CBD acid into THC and CBD vapor for inhalation. The complete 100 mg from the glass vial will be entered into the vaporizing chamber of the Volcano Medic. The vapor will be collected in a 6-L plastic balloon that, after inflation, is detached from the vaporizer and subsequently equipped with a mouthpiece for inhalation. It is our experience that the full content of the balloon is inhaled without any problems within 3-5 min.

The Bedrocan cannabis variety contains 22% THC (220 mg per gram) and less than 1%CBD. It is developed in the Netherlands out of a requirement by the Dutch Health Ministry to have a "high THC" variety available to patients. We will administer 100 mg Bedrocan that contains 22.4-mg THC and less than 1-mg CBD, twice. Bedrocan will be obtained via the Bureau voor Medicinale Cannabis (BMO), a governmental organization (VWS) that obtains cannabis from Bedrocan Int. BV in Veenendaal, The Netherlands.

Blood sampling Ten mL blood samples will be obtained on 14 occasions on each visit (total volume = 112 mL per visit) at t = 30 and 60 min after oxycodone intake and at t = 5, 20, 40, 60, 120, 180, 185, 200, 220, 240, 300 and 360 min after the first THC inhalation. From these sample, the following drugs will be measured: oxycodone, THC, THC's metabolite 11-OH-THC and cannabidiol (CBD). CBD is measured as it is expected that some minor quantities of CBD are present in Bedrocan.

Arterial blood will be collected in EDTA tubes. After blood collection the tubes will preferably be put in ice water in aluminum foiled containers, will be centrifuged within one hour for 10 minutes at 2000 G at 4 °C. The handling of samples will be done with the lights switched off. The plasma will be equally divided in 2 tubes (Brown Sarstedt) (primary and back-up sample). Plasma samples will be stored at a temperature of -80 °C and blood samples will be sent to Analytical Biochemical Laboratory (ABL) B.V., Assen, The Netherlands on dry-ice. Pharmacokinetic analysis will be performed using a validated assay. Determination of drug concentrations will be performed using liquid chromatography with tandem-mass spectrometer detection (LC-MS/MS). Analysis of the samples and acceptance criteria are indicated in ABL Standard Operating Procedure (SOP) 0251.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years,
* body mass index < 30 kg.m-2,
* able to understand the written informed consent form,
* able to communicate with the staff,
* able and willing to complete the study procedures,
* signed the informed consent form,
* deemed suitable by the investigators.

Exclusion Criteria:

* Presence or history of any medical or psychiatric disease (incl. a history of substance abuse, anxiety, or the presence of a painful syndrome such as fibromyalgia);
* Use of any medication in the three months prior to the study (incl. paracetamol or other pain killers), except for oral contraceptives (females);
* Use of more than 21 alcohol units per week;
* Use of cannabis in the 4 weeks prior to the study;
* A positive urinary drug test or a breath alcohol test at screening or on the morning of the experiment;
* Pregnancy, lactating or a positive pregnancy test on the morning of the experiment;
* Participation in another drug trial in the 60 days prior to dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The effect of inhaled THC on ventilation (Liters per minute) at an end-tidal PCO2 = 55 mmHG without and with concomitant intake of 20 mg oxycodone immediate release (IR) capsule in healthy volunteers 120 min after oxycodone intake. | 120 minutes after oxycodone intake
  As stated above

SECONDARY OUTCOMES:
Bowdle questionnaire score; | Time 0, 30, 90, 150, 210, 270, 330, 390 and 450 minutes after oxycodon or placebo administration.
  Three factors of psychedelic effects can be derived from the Bowdle questionnaire: drug high, internal perception, and external perception. Internal perception reflects inner feelings that do not correspond with the reality and is derived from questions regarding the hearing of unrealistic voices or sounds and having unrealistic thoughts and paranoid or anxious feelings. The external perception indicates a misperception of an external stimulus or change in the awareness of the subject's surroundings and is derived from questions regarding the change of body parts, the change of surroundings, the altered passing of time, the difficulty of controlling thoughts, and the change in color and sound intensity.
Pain Pressure Threshold (mN); | Time 0, 25, 55, 90, 105, 125, 145, 205, 265, 270, 285, 305, 325, 385 and 445 minutes after oxycodon or placebo administration.
  We will use the FPN 100 N Algometer (FDN 100, Wagner Instruments Inc., Greenwich, CT, USA; Rolke et al., 2005) to deliver pressure pain on a skin area of 1 cm2 between thumb and index finger. The FDN 100 has a force capacity (± accuracy) of 100 ± 2 N (10 ± 0.2 kgf) and graduation of 1 N (100 gf), respectively. A gradually increasing pressure is manually applied and the subjects are asked to indicate when the procedure becomes painful (pressure pain threshold, PPTh).
slope of the hypercapnic ventilatory response; | Time 0, 60, 120, 180, 240, 300, 360 and 420 minutes after oxycodon or placebo administration.
  Slope
plasma concentrations of THC, 11-OH-THC and oxycodone; a secondary analysis will be performed on the pharmacokinetic and pharmacodynamic data (PKPD modeling). | Time 0, 30, 60, 95, 110, 130, 150, 210, 270, 275, 290, 310, 330, 390 and 450 minutes after oxycodon or placebo administration.
  Plasma concentration
Bond & Lader questionnaire score | Time 0, 30, 90, 150, 210, 270, 330, 390 and 450 minutes after oxycodon or placebo administration.
  The Bond and Lader scales are calculated from sixteen 100 mm visual analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Monique van Velzen, Phd, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05235503/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT05235503/ICF_001.pdf